CLINICAL TRIAL: NCT04596917
Title: Music Listening as a Postanesthesia Care Unit (PACU) Nursing Intervention After Laparoscopic Radical Prostatectomy
Brief Title: Music Listening as a Postanesthesia Care Unit (PACU) Nursing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00200771
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
Keywords: music listening; Prostate Cancer; anxiety; pain management; postoperative
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized comparative study comparing two types of music listening interventions of preferred music with Spotify compared to hypnotic music with relaxation and breathing narrative
Who Masked: Participant, Care Provider, Investigator
Masking Description: PI will be working collaboratively with primary nurse. Both PI and primary nurse will maintain nursing personal protective equipment (PPE) standard of care required for the PreOp and PACU units. Prep and PACU nurses will be blinded to type of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred music listening (Experimental): Patients will be randomized to listen to music with iPod that has preferred music selections that patients can choose.
  Interventions: Behavioral: Preferred music listening
- Hypnotic music with relaxation breathing (Experimental): Patients will be randomized to listen to hypnotic music with relaxation breathing narrative.
  Interventions: Behavioral: Relaxation breathing narrative over hypnotic music listening

INTERVENTIONS:
Behavioral: Preferred music listening — The preferred music listening group will receive 15 minute patient-preferred music listening selection intervention in the Prep Room and unlimited music listening selection intervention in the PACU once cognitively ready until discharge criteria met.
  Arms: Preferred music listening
Behavioral: Relaxation breathing narrative over hypnotic music listening — The relaxation breathing group will receive the relaxation and breathing instructions over soft monotone hypnotic music in the PreOp unit before surgery and then in the PACU once cognitively ready to listen to the hypnotic music until discharge criteria met.
  Arms: Hypnotic music with relaxation breathing

SUMMARY:
A randomized comparison clinical trial will be conducted in laparoscopic radical prostatectomy patients in the Weinberg PACU at the Johns Hopkins Hospital. 50 patients will be recruited and randomly assigned by a table of random numbers to either the music listening group (n=35) or the relaxation breathing group (n=35).

DETAILED DESCRIPTION:
Hypothesis:

Laparoscopic radical prostatectomy patients who experience music listening will report decreased anxiety scores and improved pain control scores compared with patients listening to relaxation and breathing.

Null Hypothesis:

There will be no difference in reported anxiety scores and pain control scores between laparoscopic radical prostatectomy patients listening to music versus listening to relaxation and breathing instructions.

Music listening participants who meet inclusion criteria will be consented in the PreOp Unit and asked to complete the Spielberg State Trait Anxiety Inventory (STAI) questionnaire. Patient vital signs will be taken and patient will be invited to listen to music study iPod for 15 minutes prior to changing into a hospital gown.

Intervention:

The music listening group will receive the standard care and a 15 minute patient-preferred music listening selection intervention in the Prep Room and unlimited music listening selection intervention in the PACU once cognitively ready until discharge criteria met. The relaxation breathing group will receive the relaxation and breathing instructions over soft monotone music in the PACU once cognitively ready until discharge criteria met.

Results:

The experimental music listening group will reveal statistically significant decrease postanesthesia anxiety and pain, while lowering the blood pressure, heart rate and amount of opioids after laparoscopic radical prostatectomy surgery compared to the control group.

Conclusion:

The findings of the music listening intervention will provide further evidence to support the practice of music listening to decrease postanesthesia anxiety and pain, while lowering the blood pressure, heart rate and amount of opioids after laparoscopic radical prostatectomy surgery.

ELIGIBILITY:
Inclusion Criteria

* All adult male patients schedule to have a laparoscopic radical prostatectomy surgery who are ages 45 to 80 years of age
* All ethnic backgrounds
* All religions

Exclusion Criteria:

* All patients who do not speak or understand the English language to the extent that it precludes their ability to provide informed consent for the study

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men between the ages of 45 to 80 years and who are scheduled for laparoscopic radical prostatectomy surgery will be recruited.
Enrollment: 77 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety as assessed by Spielberg STAI Questionnaire | Baseline and at recovery from PACU, up to 120 minutes
  The Spielberg STAI Questionnaire has a score range of 20-80, with higher scores indicating greater anxiety.
Change in pain score | Baseline and at recovery from PACU, up to 120 minutes
  Pain will be assessed on a 0-10 scale with higher scores signifying more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Myrna E Mamaril, DNP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SW, Choi HJ. Effect of Music on Reducing Anxiety for Patients Undergoing Transrectal Ultrasound-Guided Prostate Biopsies: Randomized Prospective Trial. Urol J. 2016 Apr 16;13(2):2612-4. PMID 27085561
- [Background] Gallagher LM, Gardner V, Bates D, Mason S, Nemecek J, DiFiore JB, Bena J, Li M, Bethoux F. Impact of Music Therapy on Hospitalized Patients Post-Elective Orthopaedic Surgery: A Randomized Controlled Trial. Orthop Nurs. 2018 Mar/Apr;37(2):124-133. doi: 10.1097/NOR.0000000000000432. PMID 29570546
- [Background] Engwall M, Duppils GS. Music as a nursing intervention for postoperative pain: a systematic review. J Perianesth Nurs. 2009 Dec;24(6):370-83. doi: 10.1016/j.jopan.2009.10.013. PMID 19962104
- [Background] Barnett ML, Gray J, Zink A, Jena AB. Coupling Policymaking with Evaluation - The Case of the Opioid Crisis. N Engl J Med. 2017 Dec 14;377(24):2306-2309. doi: 10.1056/NEJMp1710014. No abstract available. PMID 29236636
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Kohler N, Friedrich M, Gansera L, Holze S, Thiel R, Roth S, Rebmann U, Stolzenburg JU, Truss MC, Fahlenkamp D, Scholz HJ, Brahler E. Psychological distress and adjustment to disease in patients before and after radical prostatectomy. Results of a prospective multi-centre study. Eur J Cancer Care (Engl). 2014 Nov;23(6):795-802. doi: 10.1111/ecc.12186. Epub 2014 Feb 13. PMID 24661440
- [Background] Liu Y, Petrini MA. Effects of music therapy on pain, anxiety, and vital signs in patients after thoracic surgery. Complement Ther Med. 2015 Oct;23(5):714-8. doi: 10.1016/j.ctim.2015.08.002. Epub 2015 Aug 4. PMID 26365452
- [Background] Maggi M, Gentilucci A, Salciccia S, Gatto A, Gentile V, Colarieti A, Von Heland M, Busetto GM, Del Giudice F, Sciarra A. Psychological impact of different primary treatments for prostate cancer: A critical analysis. Andrologia. 2019 Feb;51(1):e13157. doi: 10.1111/and.13157. Epub 2018 Oct 3. PMID 30281167
- [Background] Poulsen MJ, Coto J. Nursing Music Protocol and Postoperative Pain. Pain Manag Nurs. 2018 Apr;19(2):172-176. doi: 10.1016/j.pmn.2017.09.003. Epub 2017 Nov 16. PMID 29153918
- [Background] Miller WL, Crabtree BF. Qualitative analysis: how to begin making sense. Fam Pract Res J. 1994 Sep;14(3):289-97. PMID 7976480
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Schmid W, Rosland JH, von Hofacker S, Hunskar I, Bruvik F. Patient's and health care provider's perspectives on music therapy in palliative care - an integrative review. BMC Palliat Care. 2018 Feb 20;17(1):32. doi: 10.1186/s12904-018-0286-4. PMID 29463240
- [Background] Nishizaki T, Sumikawa K. Tunicamycin increases desensitization of junctional and extrajunctional acetylcholine receptors expressed in Xenopus oocytes by a mechanism independent of N-glycosylation blocking. Mol Pharmacol. 1992 Jul;42(1):152-6. PMID 1635551
- [Background] Bandaragoda T, Ranasinghe W, Adikari A, de Silva D, Lawrentschuk N, Alahakoon D, Persad R, Bolton D. The Patient-Reported Information Multidimensional Exploration (PRIME) Framework for Investigating Emotions and Other Factors of Prostate Cancer Patients with Low Intermediate Risk Based on Online Cancer Support Group Discussions. Ann Surg Oncol. 2018 Jun;25(6):1737-1745. doi: 10.1245/s10434-018-6372-2. Epub 2018 Feb 21. PMID 29468607